CLINICAL TRIAL: NCT00005556
Title: Retention of Bone Marrow Donors in a National Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5101; R29HL056901 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Bone Marrow Transplantation; Blood Disease
MeSH Terms: conditions — Hematologic Diseases

SUMMARY:
To identify factors that affected the National Marrow Donor Program's (NMDP) success in retention of bone marrow volunteers.

DETAILED DESCRIPTION:
BACKGROUND:

As bone marrow transplantation becomes one of the preferred treatments for life-threatening diseases of the blood, increasing numbers of patients must seek compatible marrow from unrelated donors. The low probability of finding a good patient-donor marrow match means that between one- to two-thirds of ill patients never locate a donor with perfectly compatible marrow. Furthermore, once volunteers are identified as a preliminary match for a patient, 30 to 40 percent are either unwilling or medically unable to actually donate marrow. Thus, volunteer attrition contributes significantly to the problems already inherent in finding a suitable donor candidate.

DESIGN NARRATIVE:

The study examined the relationship of volunteer characteristics and donor center factors to volunteer psychological outcomes during two critical stages in the blood testing process and to donor center rates of volunteer cooperation at these stages.

Longitudinal and cross-sectional survey data were gathered from a total of over 2,900 potential marrow donors who were at one of two critical decision points in the process leading to donation (DR-blood-typing, CT-blood-typing), and from personnel at the 100 NMDP donor centers. These data allowed the investigators to (a) describe the distribution and interrelationships between donor center structural characteristics and the strategies centers utilize for volunteer recruitment and retention, (b) determine which donor center factors (both structural and tactical) and volunteer background characteristics best predict positive volunteer-specific psychological outcomes at later typing stages, and examine and revise models of individual volunteer-specific outcomes and aggregate across-center retention rates.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-05; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galen Switzer — University of Pittsburgh

REFERENCES:
- [Background] Dew MA, Switzer GE, DiMartini AF, Matukaitis J, Fitzgerald MG, Kormos RL. Psychosocial assessments and outcomes in organ transplantation. Prog Transplant. 2000 Dec;10(4):239-59; quiz 260-1. doi: 10.1177/152692480001000408. PMID 11232552
- [Background] Switzer GE, Dew MA, Goycoolea JM, Myaskovsky L, Abress L, Confer DL. Attrition of potential bone marrow donors at two key decision points leading to donation. Transplantation. 2004 May 27;77(10):1529-34. doi: 10.1097/01.tp.0000122219.35928.d6. PMID 15239616
- [Background] Myaskovsky L, Switzer GE, Dew MA, Goycoolea JM, Confer DL, Abress L. The association of donor center characteristics with attrition from the national marrow donor registry. Transplantation. 2004 Mar 27;77(6):874-80. doi: 10.1097/01.tp.0000116394.88804.a7. PMID 15077030